CLINICAL TRIAL: NCT05217589
Title: The Influence of Different Mood States and Emotions on the Physiologic, Metabolic, and Perceptual Responses to Feeding Before Exercise
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Old Dominion University (Other)
Responsible Party: Principal Investigator, Patrick Wilson, PhD, Associate Professor of Exercise Science, Old Dominion University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 21-180
Record Dates: First submitted 2021-12-21; First posted 2022-02-01 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Other Gastrointestinal Disorders; Cramp, Abdominal
MeSH Terms: conditions — Colic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Funny/Amusing Video Clips (Experimental): Participants will watch 5-7-min video clips that are meant to be funny/amusing
  Interventions: Other: Funny/Amusing Video Clips
- Horror/Scary Video Clips (Experimental): Participants will watch 5-7-min video clips that are meant to be scary
  Interventions: Other: Horror/Scary Video Clips
- Thrilling/Suspenseful Video Clips (Experimental): Participants will watch 5-7-min video clips that are meant to be thrilling/suspenseful
  Interventions: Other: Thrilling/Suspenseful Video Clips

INTERVENTIONS:
Other: Funny/Amusing Video Clips — Participants watch 5-7 minutes of video clips that are funny/amusing in nature
  Arms: Funny/Amusing Video Clips
Other: Horror/Scary Video Clips — Participants watch 5-7 minutes of video clips that are scary in nature
  Arms: Horror/Scary Video Clips
Other: Thrilling/Suspenseful Video Clips — Participants watch 5-7 minutes of video clips that are thrilling/suspenseful in nature
  Arms: Thrilling/Suspenseful Video Clips

SUMMARY:
Many athletes anecdotally report modifying their nutritional intake before competition in order to avoid gut problems, but no studies have evaluated whether emotional state impacts tolerance to pre-exercise feeding. Therefore, this study will use movie clips (stressful, horror, and funny/amusing) to induce different mood states and emotions, which will be followed by ingestion of food before endurance running on a treadmill. In addition, metabolic and physiologic responses to mood induction will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 55 years
2. Able to run for 30 min at a moderate-to-vigorous intensity without stopping
3. No diagnosis or signs/symptoms of cardiovascular disease (CVD) or metabolic disorders
4. Currently physically active (at least 3 days/week of exercise at a moderate or higher intensity)
5. No visual or hearing impairments interfering with ability to see and hear video clips
6. No allergies to ingredients in Boost drink

Exclusion Criteria:

1. Aged <18 or >55 years
2. Unable to run for 30 min at a moderate-to-vigorous intensity without stopping
3. A diagnosis or signs/symptoms of CVD or metabolic disorders
4. Currently physically inactive (< 3 days/week of exercise at a moderate or higher intensity)
5. Visual or hearing impairments interfering with ability to see and hear video clips
6. Allergies to ingredients in Boost drink

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Total exercise gastrointestinal symptom burden | Total GI symptom burden over a 30-minute jogging/running protocol.
  The severity of several gastrointestinal symptoms will be assessed on a validated 0-10 scale. Ratings will be collected every 5 minutes during a 30-minute treadmill jogging/running test. Scores from every 5-minute collection will be summed to calculate total GI symptom scores.
Change in emotion ratings | Change in emotion ratings between immediately pre-video and immediately post-video.
  Anxiety, fear, happiness, amusement, disgust, sadness, and anger on a 0-9 Likert scale. Emotions will be assessed before watching video clips and immediately after watching video clips.

SECONDARY OUTCOMES:
Change over time in exercise heart rate | Heart rate will be measured throughout a 30-minute treadmill jogging/running test. Change over time will be evaluated using mixed ANOVA.
  Heart rate will be measured with a chest-strap (Polar) monitor.
Substrate use | Carbohydrate and fat oxidation rates will be measured during the last 5 min of a 30-minute treadmill jogging/running test.
  Carbohydrate and fat oxidation rates will be estimated from the volumes of oxygen consumption and carbon dioxide production during exercise
Feeling Scale | Ratings on the Feeling Scale will be measured at rest before watching video clips and throughout (every 5 min) a subsequent 30-minute treadmill jogging/running test.
  The Feeling Scale is a bipolar numerical rating scale ranging from -5 to +5, with descriptors of "very bad" at -5, "neutral" at 0, and "very good" at +5.
Fatigue Scale | Ratings on the Fatigue Scale will be measured at rest before watching video clips and throughout (every 5 min) a subsequent 30-minute treadmill jogging/running test.
  The Fatigue Scale is Likert-type scale that ranges from 0 (Not Fatigued at All) to 10 (Total Fatigue).
Heart rate post-video | Heart rate will be recorded immediately after videos are viewed.
  Heart rate will be measured with a chest-strap (Polar) monitor.

CONTACTS AND LOCATIONS:
Locations (1):
- Human Performance Laboratory, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided